CLINICAL TRIAL: NCT04115475
Title: New Imaging Biomarkers for Muscular Diseases - Multispectral Optoacoustic Imaging in Spinal Muscular Atrophy
Acronym: MSOT_SMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 168_19B
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Muscular Diseases; Spinal Muscular Atrophy
Keywords: Muscular Diseases, Spinal Muscular Atrophy (SMA), MSOT
MeSH Terms: conditions — Muscular Diseases; Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (HV) (Active Comparator): * Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of muscles (left and right, total 8 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: forearm flexors;
  * physical assessment/milestones: Hammersmith Infant Neurological Examination (HINE)/ expanded Hammersmith functional motor scale (HFMSE)/ The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP Intend)/ Upper Limb Module (ULM)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Spinal Muscular Atrophy (SMA) patients (Experimental): * Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of muscles (left and right, total 8 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: forearm flexors;
  * physical assessment/milestones: Hammersmith Infant Neurological Examination (HINE)/ expanded Hammersmith functional motor scale (HFMSE)/ The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP Intend)/ Upper Limb Module (ULM)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous imaging of subcellular muscle components

SUMMARY:
This study aims to refine the capability of MSOT to characterise muscle tissue and to determine non-invasive, quantitative biomarkers for the disease assessment in patients with spinal muscular atrophy (SMA) using Multispectral Optoacoustic Tomography (MSOT).

DETAILED DESCRIPTION:
SMA is an autosomal-recessive disorder, characterized by progressive muscle weakness and atrophy with an incidence of 1/10,000. The condition is caused by a homozygous deletion or mutation in the survival motor neuron 1 (SMN1), resulting in reduced expression of the survival motor neuron (SMN) protein. This leads to the degeneration of motor neurons in the spinal cord and brain stem. A nearby related gene, survival motor neuron 2 (SMN2), could partially compensate the loss of SMN1. Individuals with a higher copy number of SMN2 do in general have a milder phenotype. New therapeutic approaches, e.g. nusinersen (spinraza©), an antisense oligonucleotide medication that modulates pre-messenger RNA splicing of the survival motor neuron 2 (SMN2) gene, are promising to help the formerly incurable children. However, most clinical trials lack primary outcomes other than clinical testing. At the moment there are no prospective, quantitative biomarkers available to detect muscle atrophy at an early age, and to follow up disease progression. As a new imaging modality, optoacoustic imaging (OAI) combines benefits of optical (high contrast) and acoustic (high resolution) imaging. Multispectral optoacoustic tomography (MSOT) is therefore capable of visualizing the distribution of endogenous absorbers by initiating laser-induced thermoelastic expansion and detection of resulting pressure waves. This imaging technique enables the label-free detection and quantification of different endogenous chromophores, such as melanin, hemoglobin, deoxyhemoglobin and lipids. Previously, it was demonstrated that MSOT is capable to monitor disease severity in Crohn's disease by detecting different signal levels of hemoglobin as markers of intestinal inflammatory activity. In this study we want to refine the capability of MSOT to characterize muscle tissue and to determine a non-invasive, quantitative biomarker for the disease assessment in SMA patients from birth using MSOT.

ELIGIBILITY:
Inclusion Criteria:

* genetically proven SMA

Exclusion Criteria:

* Pregnancy
* Tattoo on skin to be examined
* For healthy volunteers only: suspected muscular disease/myopathia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Spectral profile of muscle tissue | Single time point (1 day)
  Spectral profile of muscle tissue determined by multispectral optoacoustic tomography (MSOT) of patients with spinal muscular atrophy compared to healthy volunteers units: arbitrary units (a.u.)

SECONDARY OUTCOMES:
Muscular lipid content | Single time point (1 day)
  Quantitative lipid signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA compared to healthy control Units: arbitrary units (a.u.)
Muscular collagen content | Single time point (1 day)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA compared to healthy control Units: arbitrary units (a.u.)
Muscular myo-/hemoglobin content | Single time point (1 day)
  Quantitative myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA compared to healthy control Units: arbitrary units (a.u.)
Muscular de-/oxygenated myo-/hemoglobin content | Single time point (1 day)
  Quantitative de-/oxygenated myo-/hemoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA compared to healthy control Units: arbitrary units (a.u.)
Correlation of lipid signal with clinical data (age/disease duration) | Single time point (1 day)
  Quantitative lipid signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual clinical data (disease duration/age (in month))
Correlation of collagen signal with clinical data (age/disease duration) | Single time point (1 day)
  Quantitative collagen signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual clinical data (disease duration/age (in month))
Correlation of myo-/hemoglobin signal with clinical data (age/disease duration) | Single time point (1 day)
  Quantitative myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual clinical data (disease duration/age (in month))
Correlation of de-/oxygenated myo-/hemoglobin signal with clinical data (age/disease duration) | Single time point (1 day)
  Quantitative de-/oxygenated myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual clinical data (disease duration/age (in month))
Correlation of lipid signal with physical assessment (HINE/HFMSE/CHOP INTEND/ULM) | Single time point (1 day)
  Quantitative lipid signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual physical assessment (HINE/HFMSE/CHOP INTEND/ULM)
Correlation of collagen signal with physical assessment (HINE/HFMSE/CHOP INTEND/ULM) | Single time point (1 day)
  Quantitative collagen signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual physical assessment (HINE/HFMSE/CHOP INTEND/ULM)
Correlation of myo-/hemoglobin signal with physical assessment (HINE/HFMSE/CHOP INTEND/ULM) | Single time point (1 day)
  Quantitative myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual physical assessment (HINE/HFMSE/CHOP INTEND/ULM)
Correlation of de-/oxygenated myo-/hemoglobin signal with physical assessment (HINE/HFMSE/CHOP INTEND/ULM) | Single time point (1 day)
  Quantitative de-/oxygenated myo-/hemoglobin signal (Units: arbitrary units (a.u.)) derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA correlated with individual physical assessment (HINE/HFMSE/CHOP INTEND/ULM)
Side differences of MSOT signals | Single time point (1 day)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA compared between sides Units: arbitrary units (a.u.)
Correlation of RUCT and B-Mode Ultrasound | Single time point (1 day)
  Quantitative grey scale signal derived by reflection mode ultrasound computed tomography (RUCT) correlated with grey scale B-Mode Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — University Hospital Erlangen, Department of Pediatric and Adolescent Medicine; Regina Trollmann, MD, Principal Investigator — University Hospital Erlangen, Department of Pediatric and Adolescent Medicine
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  * Individual participant data will not be available
  * Study Protocol and Statistical Analysis Plan will be available
  * The data will be available beginning 9 months and ending 36 months following article publication.
  * The data will be available to researchers who provide a methodologically sound proposal.
  * The data will be available for individual participant data meta-analysis, only.
  * Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

REFERENCES:
- [Derived] Nedoschill E, Wagner AL, Danko V, Buehler A, Raming R, Jungert J, Neurath MF, Waldner MJ, Rother U, Woelfle J, Trollmann R, Knieling F, Regensburger AP. Monitoring spinal muscular atrophy with three-dimensional optoacoustic imaging. Med. 2024 May 10;5(5):469-478.e3. doi: 10.1016/j.medj.2024.02.010. Epub 2024 Mar 25. PMID 38531362

DOCUMENTS (2):
  • Study Protocol (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04115475/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04115475/SAP_001.pdf